CLINICAL TRIAL: NCT07261436
Title: Performance Comparison of Large Language Models in TAP Block Ultrasound Interpretation: A Double-Blind Prospective Study
Brief Title: Performance Comparison of Large Language Models in TAP Block Ultrasound Interpretation
Status: Recruiting | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: SUCCESS OF LLMs in TAP BLOCK
Record Dates: First submitted 2025-11-21; First posted 2025-12-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2025-11

CONDITIONS: Artificial Intelegence
Keywords: artificial intelligence

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Gemini 2.5 Pro Evaluation — Analysis of de-identified ultrasound videos by the Gemini 2.5 Pro artificial intelligence model. The model receives standardized prompts and provides anatomical interpretation, block success assessment, and clinical suggestion outputs.
Other: ChatGPT-5.1 Evaluation — Analysis of de-identified ultrasound videos by the ChatGPT-5.1 artificial intelligence model. The model receives the same standardized questions and produces anatomical and clinical interpretations for comparison.

SUMMARY:
The goal of this study is to learn how accurately two artificial intelligence (AI) models, Gemini 2.5 Pro and ChatGPT-5.1, can interpret ultrasound videos of the Transversus Abdominis Plane (TAP) block, a regional anesthesia technique used for pain control after surgery.

The main questions this study aims to answer are:

How accurately can each AI model identify anatomical structures on TAP block ultrasound videos? Can the AI models correctly evaluate the spread of local anesthetic and determine whether the block is successful? How closely do the AI models' answers match the evaluations of expert anesthesiologists? No additional procedures will be performed on patients. TAP blocks will be done as part of routine clinical care, and the ultrasound videos will be recorded and de-identified.

Participants will not need to do anything extra for the study. Experienced anesthesiologists will review the videos and provide expert answers. The AI models will be given the same videos and asked the same questions. A second expert, who does not know which answers came from humans or AI, will compare all responses.

The results will help researchers understand whether advanced AI systems can safely support clinicians in interpreting ultrasound-guided regional anesthesia procedures and improve education and decision-making in anesthesia practice.

DETAILED DESCRIPTION:
This study aims to evaluate how two advanced artificial intelligence (AI) models, Gemini 2.5 Pro and ChatGPT-5.1, interpret ultrasound videos of Transversus Abdominis Plane (TAP) block procedures. TAP blocks are performed as part of routine clinical care by experienced anesthesiologists. The ultrasound videos recorded during these procedures serve as the data source for this study. No additional procedures or patient involvement are required beyond standard care.

Ultrasound Video Processing All ultrasound recordings will be fully de-identified by removing patient names, dates, and any other identifying information.

Gemini 2.5 Pro will receive original video files. ChatGPT-5.1 will receive high-resolution GIF segments generated from the same recordings.

Both models will be given identical structured prompts consisting of eight clinically relevant questions about anatomic structures, needle placement, local anesthetic spread, dermatomal effects, and potential safety concerns.

Expert Participation

Two anesthesiology experts will participate independently:

Expert A will review each ultrasound video and answer the same set of eight clinical questions. These answers will serve as the primary human clinical reference.

Expert B will independently evaluate all responses, those from Expert A, Gemini, and ChatGPT-5.1, after they have been anonymized and randomly ordered. Expert B will not know whether a response originated from an AI model or a human expert. Expert B will assess anatomical accuracy, clarity, clinical appropriateness, and overall content quality for each answer.

If Expert A and Expert B disagree on the interpretation or quality assessment of any response, a third expert (Expert C), who is also experienced in ultrasound-guided regional anesthesia, will independently review the relevant responses. Expert C's evaluation will be used to resolve discrepancies and establish the final consensus.

Data Collected

For each TAP block video, the following information will be recorded:

Ultrasound and procedural details. Patient demographic descriptors (age, sex, BMI, ASA classification), used only for general characterization of the sample.

AI-related performance features such as response completeness, relevance, confidence level, and response time.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-85 years
* ASA I-III physical status
* Undergoing elective surgery with a lateral TAP block performed as part of routine anesthesia care
* Complete ultrasound-guided block procedure recorded on video
* Able to provide written informed consent

Exclusion Criteria:

* Unsuccessful or incomplete TAP block procedure
* Poor-quality ultrasound video (needle tip or anesthetic spread not visible)
* Missing demographic or clinical data
* Withdrawal of consent at any time

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult surgical patients who receive a lateral Transversus Abdominis Plane (L-TAP) block as part of routine anesthesia practice during elective operations. The population consists only of patients whose block procedures are already clinically indicated and performed by experienced anesthesiologists. No additional procedures are carried out for research purposes. Ultrasound videos obtained during standard block practice are de-identified and analyzed. The study does not involve patient follow-up or any change in clinical management.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2026-01-15 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Anatomical Interpretation Accuracy | At the time of video analysis
  For each ultrasound video, the ability of both AI models (ChatGPT-5.1 and Gemini 2.5 Pro) to correctly identify key anatomical structures of the lateral TAP block (internal oblique, transversus abdominis, fascial plane, needle tip) will be evaluated. The accuracy of each model will be compared with the expert-defined reference answer.

SECONDARY OUTCOMES:
Block Success Interpretation | At the time of video analysis.
  Assessment of whether each AI model correctly determines block success based on needle placement and local anesthetic spread, compared with expert reference evaluation.
Needle Plane Evaluation | At the time of video analysis.
  Determination of whether AI models correctly assess the needle tip location and whether it is within the correct interfascial plane (IO-TA fascia), compared with the expert reference.
Dermatomal Level Prediction | At the time of video analysis.
  Comparison of each AI model's predicted dermatomal coverage (e.g., T10-T12) with the expert-provided reference dermatomal level.
Risk Awareness Assessment | At the time of video analysis.
  Evaluation of whether each AI model correctly identifies potential risks on ultrasound images (e.g., peritoneal proximity, vascular structures).
  0 = no risk awareness, 1 = partial, 2 = complete and appropriate risk identification.
Recommendation Quality | At the time of video analysis.
  Assessment of the appropriateness of each model's suggestions (e.g., need for additional injection, repositioning) based on the ultrasound appearance.
  Qualitative scoring by expert evaluator (0-10).
Agreement Between Experts | During expert evaluation phase.
  To evaluate whether Expert A and Expert B provide consistent judgments for each parameter; and to resolve discrepancies through Expert C when needed.
  Agreement / Disagreement resolved by third expert.
AI Response Time | Captured automatically during model output.
  Time required for each AI model to generate answers to the eight standardized questions.
  Seconds (continuous variable).

CONTACTS AND LOCATIONS:
Locations (1):
- Health Science University İstanbul Kanuni Sultan Süleyman Education and Training Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided